CLINICAL TRIAL: NCT00702247
Title: Allogeneic Stem Cell Transplantation for Multiple Myeloma: a Two Step Approach to Reduce Toxicity Involving High-Dose Melphalan and Autologous Stem Cell Transplant Followed by PBSC Allografting After Low-Dose TBI
Brief Title: Tandem Autologous- Nonmyeloablative Allogeneic Transplant for Newly Diagnosed Multiple Myeloma (Trapianto Tandem Autologo-Allogenico Non Mieloablativo Nel Mieloma Alla Diagnosi)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 00019702/3174
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma - Nonmyeloablative transplantation - Autologous Transplant - Graft versus myeloma; Newly diagnosed multiple myeloma; Tandem Auto-Allo Transplant; Overall survival; Event free survival; Disease response
MeSH Terms: conditions — Multiple Myeloma | interventions — Hematopoietic Stem Cell Transplantation

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplantation

SUMMARY:
To evaluate toxicity profile and efficacy of a tandem autologous-nonmyeloablative transplant approach in newly diagnose myeloma patients younger than 65 years

ELIGIBILITY:
Inclusion Criteria:

* Durie-Salmon stage IIA-IIIB multiple myeloma
* Age > 18 and ≤ 65 years
* Previously untreated myeloma
* Presence of a sibling (potential donor)
* Bilirubins < twice normal;ALAT and ASAT < four times normal
* Left ventricular ejection fraction > 40%
* Creatinine clearances > 40 mL/min
* Pulmonary dysfunction with diffusing capacity for carbon monoxide (DLCO) > 40% and/or need for continuous oxygen supplementation
* Karnofsky performance status > 60%
* Patients must give written informed consent

Exclusion Criteria:

* Age > 65 years
* Previously treated myeloma
* Absence of a sibling (genetic randomisation cannot be applied)
* Karnofsky performance status score < 60%
* HIV-infection
* Pregnancy
* Refusal to use contraceptive techniques during and for 12 months following treatment
* Patients unable to give written informed consent
* PS. Informed consent is obtained from each patient according to the Institutional Review Boards of the participating centers. The study is conducted according to the Declaration of Helsinki.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07

PRIMARY OUTCOMES:
overall survival | yearly

SECONDARY OUTCOMES:
event free survival | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Benedetto, MD, PhD, Principal Investigator — University of Torino - Italy
Locations (1):
- Università di Torino - Azienda Ospedaliera S.Giovanni Battista, Torino, Italy

REFERENCES:
- [Derived] Bruno B, Rotta M, Patriarca F, Mattei D, Allione B, Carnevale-Schianca F, Sorasio R, Rambaldi A, Casini M, Parma M, Bavaro P, Onida F, Busca A, Castagna L, Benedetti E, Iori AP, Giaccone L, Palumbo A, Corradini P, Fanin R, Maloney D, Storb R, Baldi I, Ricardi U, Boccadoro M. Nonmyeloablative allografting for newly diagnosed multiple myeloma: the experience of the Gruppo Italiano Trapianti di Midollo. Blood. 2009 Apr 2;113(14):3375-82. doi: 10.1182/blood-2008-07-167379. Epub 2008 Dec 8. PMID 19064724